CLINICAL TRIAL: NCT06054074
Title: Efficacy of a Positive Induction Through the Use of a Virtual Reality-based Program to Modify Positive Body Image Related Variables in Patients With Low Back Pain.
Brief Title: Virtual Reality-based Induction to Improve Positive Body Image in Low Back Pain Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rosa M. Baños Rivera, Full Professor, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CEIm: 30/2021; FPU20/05798 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación)
Record Dates: First submitted 2023-06-20; First posted 2023-09-26 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Chronic Low-back Pain; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Masking Description: Participants dont know the condition
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low back pain (Experimental): Participants with low back pain. They will perform the two induction procedures.
  Interventions: Behavioral: Positive Appreciation of Body Functionality Induction; Behavioral: Negative Appreciation of Body Functionality Induction

INTERVENTIONS:
Behavioral: Positive Appreciation of Body Functionality Induction — The positive induction takes place in a virtual environment of a dressing room and includes the following methods to induce positive appreciation of body functionality: 1) a narrative that aims to take the participants back to a time in the past when they held a higher positive body image. 2) A green virtual costume, representing their body at that time in the past and the positive attitude and feelings towards their body. 3) Five daily life tasks involving the use of the lower back, accompanied by auditory reminders and visual cues (green costume) to preserve the induction effect.
Behavioral: Negative Appreciation of Body Functionality Induction — The negative induction takes place in a virtual environment of a dressing room and includes the following methods to induce a lower appreciation of body functionality: 1) a narrative that aims to take the participants back to a time in the past when they held a lower positive body image. 2) A red virtual costume, representing their body at that time in the past and the negative attitude and feelings towards their body. 3) Five daily life tasks involving the use of the lower back, accompanied by auditory reminders and visual cues (red costume) to preserve the induction effect.

SUMMARY:
The aim of this study is to examine the effects of a Virtual Reality-based induction to modify positive body image in individuals with low back pain.

Participants will receive both a positive and a negative induction of the appreciation of body functionality. This induction consists of an elaborated narrative to increase/decrease the appreciation of functionality. In addition, each induction includes a virtual costume representing their body's strengths or weaknesses to enrich the induction. After both induction procedures, participants will perform activities of daily living involving the use of the lumbar region in virtual reality. Subsequently, the different variables of interest will be assessed before and after each induction.

Researchers will analyze changes in the variables of interest after induction procedures compared to baseline.

DETAILED DESCRIPTION:
The aim of this study is to examine the effects of a Virtual Reality-based induction to modify positive body image in individuals with low back pain.

Firstly, improvement in the study variables is expected after the positive induction. Secondly, the opposite results are expected after negative induction. Thirdly, a greater change is expected in the group of patients with low back pain.

The whole study is conducted in one single 1-hour session. First, participants will be screened to check eligibility inclusion/exclusion criteria. Second, eligible participants will complete baseline measures. Third, participants will be exposed to both induction procedures, counterbalancing the order. At the end of each induction, they will have to perform different virtual reality-based tasks of daily life that involve the use of the lumbar region, such as placing books on a bookshelf, throwing objects into a trash can or painting a wall. Fourth, state measures will be applied to assess the change in the study variables.

The study will be conducted following the principles stated in the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with low back pain.

Exclusion Criteria:

Meeting any of the following medical conditions:

* Spinal tumor, infection or fracture
* Systemic disease (autoimmune, infectious, vascular, endocrine, metabolic...)
* Fibromyalgia
* Cauda equina syndrome
* History of spinal surgery
* Musculoskeletal injury of lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Appreciation of Body Functionality: Baseline | The whole study is conducted in a single experimental session: Immediately before induction procedures.
  Baseline measure of Functionality Appreciation Scale (FAS). The scores range from 1 to 5, where higher scores indicates higher levels of appreciation of body functionality.
Appreciation of Body Functionality: Post positive induction procedure | The whole study is conducted in a single experimental session: Immediately after positive induction procedure.
  Post positive induction measure of FAS. The scores range from 1 to 5, where higher scores indicates higher levels of appreciation of body functionality.
Appreciation of Body Functionality: Post negative induction procedure | The whole study is conducted in a single experimental session: Immediately after negative induction procedure.
  Post negative induction measure of FAS. The scores range from 1 to 5, where higher scores indicates higher levels of appreciation of body functionality.
Body Awareness: Body Trusting; Baseline | The whole study is conducted in a single experimental session: Immediately before induction procedures.
  Baseline measure of "Trusting" subscale from Multidimensional Assessment of Interoceptive Awareness-2 (MAIA-2). The scores range from 0 to 5, where higher scores indicate a higher level of trust in one's own body.
Body Awareness: Body Trusting; Post positive induction procedure | The whole study is conducted in a single experimental session: Immediately after positive induction procedure.
  Post positive induction measure of "Trusting" subscale from MAIA-2. The scores range from 0 to 5, where higher scores indicate a higher level of trust in one's own body.
Body Awareness: Body Trusting; Post negative induction procedure | The whole study is conducted in a single experimental session: Immediately after negative induction procedure.
  Post negative induction measure of "Trusting" subscale from MAIA-2. The scores range from 0 to 5, where higher scores indicate a higher level of trust in one's own body.
Positive Embodiment: Positive Body Connection and Comfort (PBCC); Baseline | The whole study is conducted in a single experimental session: Immediately before induction procedures.
  Baseline measure of PBCC subscale from Experience of Embodiment Scale (EES). The scores range from 1 to 5, where higher scores indicates a more positive experience of embodiment.
Positive Embodiment: Positive Body Connection and Comfort (PBCC); Post positive induction procedure | The whole study is conducted in a single experimental session: Immediately after positive induction procedure.
  Post positive induction measure of PBCC subscale from EES. The scores range from 1 to 5, where higher scores indicates a more positive experience of embodiment.
Positive Embodiment: Positive Body Connection and Comfort (PBCC); Post negative induction procedure | The whole study is conducted in a single experimental session: Immediately after negative induction procedure.
  Post negative induction measure of PBCC subscale from EES. The scores range from 1 to 5, where higher scores indicates a more positive experience of embodiment.
Attitudes or Feelings towards One's Own Body; Baseline | The whole study is conducted in a single experimental session: Immediately before the induction procedures and immediately after the first applied induction procedure.
  Baseline measure of a semantic differential developed to assess attitudes and feelings towards one's own body. The scores range from 0 to 10, with higher scores representing a more positive evaluation of the one's own body.
Attitudes or Feelings towards One's Own Body; Post first induction procedure | The whole study is conducted in a single experimental session: Immediately before the first induction procedure.
  Post first induction procedure measure of a semantic differential developed to assess attitudes and feelings towards one's own body. The scores range from 0 to 10, with higher scores representing a more positive evaluation of the one's own body.

SECONDARY OUTCOMES:
Pain intensity: Baseline | The whole study is conducted in a single experimental session: Immediately before the induction procedures.
  Baseline measure of pain (numerical rating scale). The scores ranges to 0: "no pain" to 10: "maximum pain".
Pain intensity: Post positive induction procedure | The whole study is conducted in a single experimental session: Immediately after positive induction procedure.
  Post positive induction measure of pain (numerical rating scale). The scores ranges to 0: "no pain" to 10: "maximum pain".
Pain intensity: Post negative induction procedure | The whole study is conducted in a single experimental session: Immediately after negative induction procedure.
  Post negative induction measure of pain (numerical rating scale). The scores ranges to 0: "no pain" to 10: "maximum pain".
Fear of movement; Post positive induction procedure | The whole study is conducted in a single experimental session: Immediately after the positive induction procedure.
  Post positive induction measure of fear of movement with a single item (numerical rating scale); ranging from 0: " No fear" to 10: "maximum fear".
Fear of movement; Post negative induction procedure | The whole study is conducted in a single experimental session: Immediately after the negative induction procedure.
  Post negative induction measure of fear of movement with a single item (numerical rating scale); ranging from 0: " No fear" to 10: "maximum fear".
Task difficulty; Post positive induction procedure | The whole study is conducted in a single experimental session: Immediately after the positive induction procedure.
  Post positive induction measure of task difficulty with a single item (numerical rating scale); ranging from 0: "very easy" to 10: "very hard".
Task difficulty; Post negative induction procedure | The whole study is conducted in a single experimental session: Immediately after the negative induction procedure.
  Post negative induction measure of task difficulty with a single item (numerical rating scale); ranging from 0: "very easy" to 10: "very hard".

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Baños, PhD, Principal Investigator — University of Valencia
Locations (1):
- Arnau de Vilanova Hospital, Valencia, Spain

REFERENCES:
- [Background] Alleva JM, Tylka TL, Kroon Van Diest AM. The Functionality Appreciation Scale (FAS): Development and psychometric evaluation in U.S. community women and men. Body Image. 2017 Dec;23:28-44. doi: 10.1016/j.bodyim.2017.07.008. Epub 2017 Aug 17. PMID 28822275
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Piran N, Teall TL, Counsell A. The experience of embodiment scale: Development and psychometric evaluation. Body Image. 2020 Sep;34:117-134. doi: 10.1016/j.bodyim.2020.05.007. Epub 2020 Jun 14. PMID 32554242